CLINICAL TRIAL: NCT00064558
Title: Genetic Determinants of Sudden Cardiac Death
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christine M. Albert, MD, MPH, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 1228; R01HL068070 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-10 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Death, Sudden, Cardiac; Ventricular Arrhythmia; Arrhythmia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Death, Sudden, Cardiac; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
To evaluate whether genetic variation in selected candidate genes is associated with risk of sudden cardiac death in the general population.

DETAILED DESCRIPTION:
BACKGROUND Sudden cardiac death (SCD) affects 400,000 individuals each year in the U.S. alone. Over half have no evidence of heart disease prior to death, and our ability to identify those at risk and, therefore prevent SCD, is poor. Mutations in cardiac ion channel genes including SCN5A, KCNQ1, KCNH2, KCNE1, KCNE2 and RyR2 have been implicated in monogenic traits with high risk of SCD, such as the long-QT, Brugada, sudden infant death syndrome (SIDS), and catecholaminergic polymorphic ventricular tachycardia. Alterations in ion channel function can result in life-threatening ventricular arrhythmias in diverse disease states. Therefore, sequence variants in these genes that alter function or transcription of these ion channels may confer a predisposition to ventricular arrhythmia and SCD in broader populations.

DESIGN NARRATIVE This research program proposes to determine if sequence variants in the above and other candidate genes are associated with an increased risk of SCD in apparently-healthy populations. Cases of SCD will be assembled from 5 NIH-funded prospective cohorts with a total of 106,314 individuals with existent blood samples. All cohorts are exceptionally well-characterized with respect to environmental exposures and have collected medical records on cardiovascular endpoints. We will characterize all coding sequence variation and selected non-coding sequence variation among 100 cases and controls from these cohorts for the 6 genes. We will then employ a nested case-control design and conditional logistic regression to test for associations between haplotypes (haplotype tag SNPs) in both coding and non-coding regions of candidate genes and SCD risk. We will also test directly for associations between single loci that may have functional significance and SCD risk. An estimated 600 cases of well-documented SCD will be confirmed over the first 3 years of the grant period, and these cases will be matched on age, sex, ethnicity, and geographic location to two control subjects from the same cohort. In addition, based upon known sex difference in the phenotypic expression of the candidate genes in the primary arrhythmic disorders, we will specifically examine sex difference in the risk of SCD associated with sequence variation in these genes. The findings generated will have substantial implications for our understanding of the SCD syndrome and risk stratification in the general population.

ELIGIBILITY:
No eligibility criteria.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants previously enrolled in the Physicians' Health Study I (Protocol 1999-P-001468), Physicians' Health Study II (Protocols 1999-P-003315, 1999-P-003318), Nurses' Health Study (Protocols 1999-P-01114, 1999-P-010982), Women's Health Study (Protocols 1999-P-001304, 1999-P-001478), Women's Antioxidant Cardiovascular Study (Protocols 1999-P-001364, 1999-P-001611), and Health Professional Health Study approved through the Harvard School of Public Health IRB (Protocols 0007PROC, 0103STOR).
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2003-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
sequence variation | Ongoing
  To determine if sequence variants in SCN5A, KVLQT1, HERG, KCNE1, KCNE2, and RyR2 genes and other candidate genes are associated with an increased risk of SCD in broader populations.

SECONDARY OUTCOMES:
Single loci and SCD risk | Ongoing
  To test directly for associations between single loci that may have functional significance and SCD risk.

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Albert, M.D., M.P.H., Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No